CLINICAL TRIAL: NCT02882997
Title: A Virtual Environment for Post-Stroke Upper Extremity Rehabilitation
Brief Title: An Interactive Computer Game, Called Duck Duck Punch, for Stroke Rehabilitation at Home and in a Rehabilitation Clinic
Acronym: DDPHme/Hsp
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Principal Investigator, Michelle Woodbury, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00029185
Record Dates: First submitted 2016-08-05; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duck Duck Punch (Experimental): Community dwelling stroke survivors: Stroke survivors will install an interactive computer game in their home. Subjects will be instructed to play the computer game "as much as you want to every day for 7 days." Inpatient stroke patients: The interactive computer game will be installed at a local inpatient stroke rehabilitation hospital. Subjects will be instructed to "play this game as much as you want to during non-therapy hours (evenings and weekends) over the next 7 days."
  Interventions: Behavioral: an interactive computer game
- Standard activities (Active Comparator): Community dwelling stroke survivors: Subjects will receive a hard-copy handout of an arm home exercise program and given the instructions to "do these exercises as many times as you can daily." Inpatient stroke patients: Subjects will be encouraged to participate in standard evening/weekend recreational activities and to "remember to use the paretic arm as much as you can."
  Interventions: Behavioral: standard activities

INTERVENTIONS:
Behavioral: an interactive computer game — Duck Duck Punch is an interactive computer game designed to elicit repetitive practice of paretic arm movements in stroke patients.
  Arms: Duck Duck Punch
Behavioral: standard activities — For community dwelling stroke survivors this is a hard copy, written/illustrated home exercise program for the paretic arm. For inpatient stroke patients this is standard recreational activities organized by the facility during non therapy hours (evenings and weekends).
  Arms: Standard activities

SUMMARY:
This study will determine the feasibility of using an interactive computer game to elicit repetitive practice of paretic arm movements in the homes of community dwelling stroke survivors and during non-therapy hours at an inpatient stroke rehabilitation hospital.

DETAILED DESCRIPTION:
More than 75% of the 800,000 people who annually suffer stroke exhibit persistent arm/hand hemiparesis restricting independence thus burdening caregivers. Arm motor skill can recover if the rehabilitation program provides an adequate "dose" of repetitive movement practice. However, the vast majority of stroke survivors lack the proper practice-dose because the duration of inpatient stroke rehabilitation is limited by cost, or residence in medically underserved rural settings. To meet the pressing need for innovative cost-effective rehabilitation options, the investigators developed, tested and licensed a prototype virtual environment (VE) for post-stroke arm rehabilitation. Its custom built design motivates extended practice of specific arm motor skills known to improve quality of life. Excitingly, practice sessions do not require direct therapist supervision. Published pilot data demonstrated improved real-world arm movement after VE training. These promising initial results led to software upgrades that will now enable installation and testing in the primary markets for this technology; stroke rehabilitation hospitals, and patients' homes. The overall goal for this small pilot study is to test the feasibility of self-directed VE practice in these settings measured by movement repetitions and motor skill improvement. To that end, this project will address the following Specific Aims (1) Determine the number of daily movement repetitions and treatment effect achieved by inpatients in a stroke rehabilitation hospital who self-direct VE practice sessions during non-therapy hours (evenings, weekends) compared to standard evening activities; and (2) Determine the number of daily movement repetitions and treatment effect achieved by in-home stroke survivors who self-direct daily VE practice sessions compared to a group of in-home survivors with a standard self-directed exercise program.

ELIGIBILITY:
Inclusion Criteria:

* experienced uni-hemispheric ischemic or hemorrhagic stroke
* exhibit voluntarily shoulder flexion (affected UE) ≥20° with simultaneous elbow extension ≥10°. We reason that persons at this motor ability level have enough residual arm activation to engage in VE training
* passive range of motion in affected shoulder and elbow and within 20 degrees of normal values

Additional inclusion criteria for community dwelling stroke survivors

* live at home
* no current rehabilitation therapy
* live within a 60 minute drive of the university

Additional inclusion criteria for inpatient stroke patients

* medically stable
* expected to remain in the hospital for the next 7 days
* able to sit in a chair for 60 minutes without difficulty

Exclusion Criteria:

* lesion in brainstem or cerebellum
* presence of other neurological disease that may impair motor skills (e.g., Parkinson's Disease)
* pain in the paretic arm that would interfere with movement
* unable to understand and follow 3-step directions
* orthopedic condition or impaired corrected vision that would interfere with reaching.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Paretic arm use | 1 year
  The amount of paretic arm use will be measured by wrist worn accelerometers. Subjects will be shown how to don/doff wristwatch sized triaxial Actigraph accelerometers (GT3X+ Activity Monitor; ActiGraph LLC) by securing a Velcro band on the dorsal aspect of each wrist proximal to the wrist joint. Subjects will be instructed to don the accelerometers each time they engaged in either the computer game or standard activity and wear them only for the duration of the activity. The accelerometers will be stored in a box during other times. Accelerometry data will be recorded in 1 minute epochs as the number of arm activity counts. At the final study evaluation session, data will be used to create a ratio of paretic to non-paretic arm activity counts. A value of 1 will indicate bilateral arm use, a value higher than 1 will indicate that the paretic arm was used more than the non-paretic arm, and a value less than 1 will indicate that the paretic arm was used less than the non-paretic arm.

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment | up to 7 days
  a 33-item measure of arm impairment testing the subject's ability to achieve various postures with the paretic arm and hand, scored on a 3 point ordinal rating scale with higher scores indicating less motor impairment.
Wolf Motor Function Test | up to 7 days
  A 15-item evaluation of paretic arm motor function, testing the amount of time required for a subject to use the paretic arm to accomplish various functional tasks.
Stroke Impact Scale - Hand subtest | up to 7 days
  A 5-item evaluation of patient self-reported level of difficulty using the paretic hand to perform various functional activities at home. Items are rated on a 4 point ordinal scale so that higher numbers indicate less difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Woodbury, PhD, OTR/L, Principal Investigator — Medical University of South Carolina
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Woodbury ML, Anderson K, Finetto C, Fortune A, Dellenbach B, Grattan E, Hutchison S. Matching Task Difficulty to Patient Ability During Task Practice Improves Upper Extremity Motor Skill After Stroke: A Proof-of-Concept Study. Arch Phys Med Rehabil. 2016 Nov;97(11):1863-1871. doi: 10.1016/j.apmr.2016.03.022. Epub 2016 Apr 23. PMID 27117385
- See also: A paper presented at a conference on the initial development of the interactive computer game. — http://ieeexplore.ieee.org/xpl/articleDetails.jsp?reload=true&arnumber=6550196